CLINICAL TRIAL: NCT02704559
Title: Study to Explore Drug-drug Interactions Between DWC20155 and DWC20156 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1366001
Record Dates: First submitted 2016-02-27; First posted 2016-03-10 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy

ARMS (2):
- Study effect of DWC20156 on DWC20155 PK (Experimental): To study effect of DWC20156 on DWC20155 PK
  Interventions: Drug: DWC20156
- Study effect of DWC20155 on DWC20156 PK (Experimental): To study effect of DWC20155 on DWC20156 PK
  Interventions: Drug: DWC20155

INTERVENTIONS:
Drug: DWC20155
  Arms: Study effect of DWC20155 on DWC20156 PK
Drug: DWC20156
  Arms: Study effect of DWC20156 on DWC20155 PK

SUMMARY:
A randomized, open-label, oral dose, crossover study to explore drug-drug interactions between DWC20155 and DWC20156 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Accepts healthy volunteers.

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0~24hr
Area under the plasma concentration versus time curve (AUC) | 0~24h

CONTACTS AND LOCATIONS:
Locations (1):
- Busan Paik Hospital, Busan, South Korea